CLINICAL TRIAL: NCT06104514
Title: Safety and Efficacy of Sofwave Treatment to Lift the Upper Lip and Improve the Peri-Oral Rhytids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sofwave Medical LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sofwave20
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Rhytides; Wrinkle
Keywords: upper lip, peri-oral, philtral
MeSH Terms: conditions — Lymphoid Interstitial Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Lift the upper lip and improve the peri-oral rhytids (Experimental)
  Interventions: Device: Sofwave

INTERVENTIONS:
Device: Sofwave — The Sofwave System, comprised of an applicator and a console, generates high intensity, non-focused ultrasonic energy which can be delivered percutaneously to tissues.
  Other Names: SUPERB

SUMMARY:
Open-label, non-randomized, prospective, multi-center, self-controlled

DETAILED DESCRIPTION:
Patients will receive 2 monthly treatments with the SofWave system and will be followed up twice: at 4 weeks and 12 weeks after last treatment (FU1-FU2).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female and male subjects between the ages 35-80.
2. Desire to improve the peri-oral appearance, decrease the distance between the nose and the upper lip (Philtral column length) and/or reduce the peri-oral rhytids.
3. Philtral column height>15mm or/and has moderate severe perioral rhytids.
4. Subject agrees to maintain a stable weight (i.e., within 5% of total body weight) by not making any major changes in their diet or exercise routine during the study.
5. Able and willing to comply with all visits, treatments and evaluation schedules and requirements.
6. Able to understand and provide written Informed Consent.
7. Willing to have photographs of the treated areas. Agree for de-identified study images to be used in evaluations, publications and presentations.
8. Agree not to undergo any other facial treatments for a period of 3 months following SofWave treatments.
9. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment.

Exclusion Criteria:

1. Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breast feeding.
2. Current smoker or has history of heavy smoking (25 cigarettes per day or more) in past 10 years.
3. Melanoma active malignancy or history of malignancy in the past 5 years.
4. Any other non-melanoma malignancy active malignancy or history of malignancy in the past 5 years within the intended to treat area.
5. Previous chemotherapy treatments.
6. Suffering from significant concurrent illness, such as cardiac disorders, diabetes (type I or II), lupus, porphyria, or pertinent neurological disorders (i.e. any disease state that in the opinion of the investigator may interfere with the anesthesia, treatment, or healing process).
7. History of chronic drug or alcohol abuse
8. History of Epileptic seizures.
9. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
10. Suffering from hormonal imbalance, whether related to thyroid, pituitary, or androgen.
11. History of significant lymphatic drainage problems within the facial areas.
12. History of epidermal or dermal disorders (particularly involving collagen or microvascularity), including collagen vascular disease or vasculitic disorders.
13. Excessive subcutaneous fat on the face.
14. Taking Isotretinoin or other oral retinoid within the past 6 months; taking anti-coagulant within the past 2 weeks
15. Currently taking or has taken diet pills or weight control supplements within the past month.
16. Non-stable weight ( ±5%) within the past month.
17. Medical disorder that may hinder the wound healing or immune response (such as blood disorder, inflammatory disease, etc.)
18. Known allergy to Lidocaine, Tetracaine, Xylocaine, Epinephrine or antibiotics.
19. Skin disorders (skin systematic or local infections or rashes, extensive scarring, psoriasis, etc.) in the treatment area.
20. Severe solar elastosis at the intended to treat area.
21. Tattoo or former tattoo at or near treatment area.
22. Tendency for Melasma inflammation.
23. Significant scarring, atrophic scars in the area to be treated, or has a history of atrophic scars or keloids or prone to bruising.
24. Surgical or traumatic scar in the intended to treat area.
25. Presence of a metal stent or implant in the facial area (e.g. braces; dental implants are not excluded).
26. History of cosmetic treatments in the facial area to be treated, including blepharoplasty, direct specific forehead lift and facial skin-tightening procedure within the 6 months;injectable (Botox or fillers) of any type within the 12 months; ablative or non-ablative resurfacing/rejuvenation laser treatment or light treatment within the past 6 months, dermabrasion or deep facial peels within the past 12 months; facelift or neck lift within the past 12 months.
27. Currently enrolled in a clinical study of any other unapproved investigational drug or device.
28. As per the investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Rate of improvement in the appearance of upper lip and peri-oral rhytids | 12 weeks post last treatment
  Study will be considered a success if more than 50% of the subjects will have an improvement according to investigators' assessments of pre- and post Treatment 2D images

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Premier Plastic Surgery, Palo Alto, California
  - Cosmetic Laser Dermatology, San Diego, California
  - Advanced dermatoloy, Lincolnshire, Illinois
  - Aesthetic Revolution Las Vegas, Las Vegas, Nevada
  - New Jersey Plastic Surgeon, Montclair, New Jersey
  - UnionDerm, New York, New York